CLINICAL TRIAL: NCT00939861
Title: Study Comparing Laparoscopy Versus Laparotomy in the Treatment of Colorectal Endometriosis
Brief Title: Laparoscopy Versus Laparotomy for Colorectal Endometriosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tenon Hospital, Paris (Other)
Responsible Party: Emile Daraï, Departement of Obstetrics and Gynecology, Tenon Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13072009
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Endometriosis
Keywords: colorectal endometriosis, laparoscopy, laparotomy; gynecologic and digestive symptoms; quality of life (SF-36 questionnaire); morbidity; fertility
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): laparoscopy
  Interventions: Procedure: laparoscopy
- 2 (Experimental): laparotomy
  Interventions: Procedure: laparotomy

INTERVENTIONS:
Procedure: laparoscopy — colorectal resection
  Arms: 1
Procedure: laparotomy — colorectal resection
  Arms: 2

SUMMARY:
Study hypothesis: equivalency of laparoscopic compared to laparotomic colorectal resection for endometriosis on digestive, gynaecologic, general symptoms and quality of life. Morbidity and fertility outcomes will also be evaluated.Primary purpose of the protocol is the evaluation of dyschesia.

DETAILED DESCRIPTION:
For all patients, colorectal endometriosis will be confirmed preoperatively by clinical examination, transvaginal sonography, rectal endoscopic sonography and magnetic resonance imaging.Among patients with an indication of surgery, the intensity of dyschesia and other gynecological or digestive disorders will be evaluated pre-operatively using a visual analogue scale. Quality of life will be assessed using the SF-36 questionnaire. The allocation of the surgical route will be conducted by lottery the day before surgery. Patients will be reviewed postoperatively at 1 month and a new assessment of symptoms will be made at 6 months. The duration of the study will be 7 months for the patient and 24 months in total.If considering the two surgical routes as equivalent, with a delta score (after-before surgery) = ±2, standard deviation = 1.55, risk α=2.5%, risk β=10%, and taking into account that prevalence of dyschesia in the study population is 63%, 52 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* patients with colorectal endometriosis
* patients affiliated to the French Health Care system
* patients having signed the inform consent.
* patients who can speak and read French

Exclusion Criteria:

* patients with prior colorectal surgery
* patients with a contraindication to laparoscopy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dyschesia at 6 months using a visual analogue scale | at 6 months

SECONDARY OUTCOMES:
Evaluation of gynaecologic symptoms (dysmenorrhea, dyspareunia), digestive symptoms (diarrhea, constipation , intestinal cramps) and general symptoms (asthenia, back pain) at 6 months using visual analogue scale | at 6 months
Evaluation of quality of life at 6 months using SF-36 questionnaire | at 6 months
Morbidity | During 6 months
Postoperative fertility | during the study

CONTACTS AND LOCATIONS:
Overall Officials: emile Daraï, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Tenon Hospital, Departement of Obstetrics and Gynecology, Paris, Paris, France

REFERENCES:
- [Derived] Touboul C, Ballester M, Dubernard G, Zilberman S, Thomin A, Darai E. Long-term symptoms, quality of life, and fertility after colorectal resection for endometriosis: extended analysis of a randomized controlled trial comparing laparoscopically assisted to open surgery. Surg Endosc. 2015 Jul;29(7):1879-87. doi: 10.1007/s00464-014-3880-4. Epub 2014 Oct 8. PMID 25294552